CLINICAL TRIAL: NCT03702023
Title: Oral Acetaminophen Use for Pain Reduction in Electrophysiology Procedures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ascension Health (Industry)
Responsible Party: Principal Investigator, Andrew Hinojos, Cardiology Fellow, Ascension Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Acetaminophen in EP procedures
Record Dates: First submitted 2018-08-23; First posted 2018-10-10 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Post Electrophysiology Procedure Pain
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention Group (Active Comparator): Patients in the intervention group with receive the study medication 1000mg acetaminophen orally one time prior to their scheduled electrophysiology procedure.
  Interventions: Drug: Acetaminophen
- Placebo Oral Tablet (Placebo Comparator): Patients in the control group will receive a placebo orally one time prior to their scheduled electrophysiology procedure.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Acetaminophen — Intervention group will receive 1000 mg of acetaminophen
  Other Names: Tylenol
  Arms: Intervention Group
Drug: Placebo Oral Tablet — Control group will be given a placebo capsule.
  Other Names: Placebo
  Arms: Placebo Oral Tablet

SUMMARY:
The investigators are purposing a study to evaluate the use of acetaminophen given prior to an electrophysiology procedure and post procedural pain control.

DETAILED DESCRIPTION:
Atrial arrhythmias are very common and widespread. Recent reports suggest that 9% of patients over the age of 65 currently have atrial fibrillation. In individuals of European descent the lifetime risk of atrial fibrillation is as high as 26%. Atrial fibrillation carries significant risk of complications including: a fivefold increase in risk of stroke, a threefold risk of heart failure, a twofold risk of dementia and a twofold risk of mortality. As treatment options continue to evolve, the use of catheter ablation procedures are becoming increasingly common within the United States. Currently, ablation has a class 1A recommendation for patients with symptomatic paroxysmal atrial fibrillation refractory or intolerant to at least one class I or class III antiarrhythmic medication and a class 2B indication before initiation of antiarrhythmic drug therapy. One of the known complications of catheter ablation procedures is pain following the procedure. Severe pain has been reported in up to 55% of patients undergoing ablation procedures. IV acetaminophen has been proven to be effective at controlling pain in post intra-abdominal surgery, however, its use is limited due to the cost of this medication. Other studies have suggested that there is no clear indication for IV over oral acetaminophen in patients who are able to take oral. Empirically the investigators have seen patients complaining of pain after all electrophysiology procedures, not limited to just ablation procedures. To the best of the knowledge of the investigational team, at this time, no studies have looked at using oral pre-procedural acetaminophen to assist with pain control following electrophysiology procedures. The investigators are looking to perform a randomized, double blind, placebo controlled study to evaluate the use of pre-procedural oral acetaminophen to help control post procedural pain.

ELIGIBILITY:
Inclusion Criteria:

* Age: Over 18
* Weight: Greater than 50kg
* Scheduled for an EP procedure
* Be able to take oral medications
* Provide signed written informed consent

Exclusion Criteria:

* Have chronic pain requiring the use of chronic pain medications including narcotic pain medications or chronic acetaminophen use greater than seven consecutive days prior to the procedure
* Known hypersensitivity to acetaminophen
* Known or suspected history of alcohol or drug abuse/dependence within the previous 2 years
* Known impaired liver function
* Active pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-02-08 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale measurement of pain in response to electrophysiology procedures and change in pain over time. | The patients pain will be recorded prior to the procedure and then every one hour post procedure for four hours. Pain will then be recorded every four hours for a total of 24 hours or patient discharge from the hospital whichever comes first.
  A standard 0-10 numerical rating scale of pain (0=no pain, 10 = the worst possible pain) will be subjectively reported to nursing staff and recorded.

SECONDARY OUTCOMES:
Additional Pain Medication | We will monitor the patients for additional doses of pain medication from the time their procedure is completed and the following 24 hours.
  Duration of time from the start of the procedure until the next dose of pain medication is provided. We will be monitoring the type and dose of pain medication provided.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Taipale, D.O., Principal Investigator — Ascension Health
Locations (1):
- Ascension Genesys Hospital, Grand Blanc, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No plans at this time to share IPD with other researchers

REFERENCES:
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; ACC/AHA Task Force Members. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines and the Heart Rhythm Society. Circulation. 2014 Dec 2;130(23):2071-104. doi: 10.1161/CIR.0000000000000040. Epub 2014 Mar 28. No abstract available. PMID 24682348
- [Background] Bode K, Breithardt OA, Kreuzhuber M, Mende M, Sommer P, Richter S, Doering M, Dinov B, Rolf S, Arya A, Dagres N, Hindricks G, Bollmann A. Patient discomfort following catheter ablation and rhythm device surgery. Europace. 2015 Jul;17(7):1129-35. doi: 10.1093/europace/euu325. Epub 2014 Dec 8. PMID 25488958
- [Background] Wininger SJ, Miller H, Minkowitz HS, Royal MA, Ang RY, Breitmeyer JB, Singla NK. A randomized, double-blind, placebo-controlled, multicenter, repeat-dose study of two intravenous acetaminophen dosing regimens for the treatment of pain after abdominal laparoscopic surgery. Clin Ther. 2010 Dec;32(14):2348-69. doi: 10.1016/j.clinthera.2010.12.011. PMID 21353105
- [Background] Jibril F, Sharaby S, Mohamed A, Wilby KJ. Intravenous versus Oral Acetaminophen for Pain: Systematic Review of Current Evidence to Support Clinical Decision-Making. Can J Hosp Pharm. 2015 May-Jun;68(3):238-47. doi: 10.4212/cjhp.v68i3.1458. PMID 26157186